CLINICAL TRIAL: NCT07341113
Title: Effects of Body Position on Ventilation and Perfusion Distribution in Obese and Non-Obese Healthy Volunteers Assessed by Electrical Impedance Tomography
Brief Title: Positional Effects on Lung Ventilation and Perfusion in Obesity
Status: Active, not recruiting | Type: Observational
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025.510.IRB2.232
Record Dates: First submitted 2025-12-15; First posted 2026-01-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Obesity (Disorder); Ventilation Homogeneity; Perfusion; Ventilation Perfusion Mismatch; Position Differences; Electrical Impedance Tomography (EIT)
Keywords: obesity; ventilation perfusion; electrical impedance tomography; body positions
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-obese group: Non-obese healthy individuals with BMI between 18.5 - 25 kg/m²
  Interventions: Other: Standardized body positioning
- Obese group: Obese healthy individuals with BMI between 30 - 40 kg/m²
  Interventions: Other: Standardized body positioning

INTERVENTIONS:
Other: Standardized body positioning — Standardized changes in body position (supine, Trendelenburg, prone, and lateral positions) performed solely for physiologic assessment of ventilation and perfusion using electrical impedance tomography. This does not constitute a therapeutic or preventive intervention.

SUMMARY:
Electrical Impedance Tomography (EIT) is a non-invasive, bedside monitoring tool that provides real-time information on regional ventilation and perfusion. In particular, EIT has the potential to guide individualized mechanical ventilation in obese patients by revealing how gravitational and positional factors alter regional lung behavior. Assessing the effects of different horizontal positions on both ventilation and perfusion may help optimize respiratory management strategies tailored to body habitus. By comparing obese and non-obese healthy participants across different positions, this study aims to provide novel insights into the postural effects on lung aeration and perfusion distribution, and to highlight the role of EIT in tailoring individualized ventilation strategies.

DETAILED DESCRIPTION:
This will be a observational, physiological study involving healthy volunteers divided into two groups: Obese group (BMI 30 - 40 kg/m²) and non-obese group (BMI 18.5 - 24.9 kg/m²). Each participant will serve as their own control across body positions. Baseline measurements will be obtained in upright sitting, followed by randomized order of supine, Trendelenburg (30°), prone, left lateral, and right lateral. Participants' demographic and anthropometric data, including height, weight, chest circumference, waist circumference, and hip circumference, will be recorded. Medical history, current medication use, smoking status, and cumulative smoking exposure (pack-years) will be documented.

Electrical Impedance Tomography (EIT) measurements will be performed using the Infivision ET1000 device. All study procedures will take place in a private room within the General Intensive Care Unit of Koç University Hospital, with privacy ensured throughout the protocol. After removal of upper body clothing, an appropriately sized EIT belt, selected according to chest circumference, will be positioned circumferentially around the thorax at the level of the axillae. A pulse oximetry probe will be applied, and continuous monitoring of heart rate and peripheral oxygen saturation will be maintained during all measurements.

Following a 5-minute stabilization period in the upright sitting position, baseline EIT measurements will be obtained. The following parameters will be recorded: percentage of ventral ventilation, percentage of dorsal ventilation, percentage of ventral perfusion, percentage of dorsal perfusion, Match Index (MI), Dead Space Index (DI), Shunt Index (SI), Global Inhomogeneity Index (GI), and Center of Ventilation (CoV). To minimize potential carry-over effects, the sequence of positions will be randomized individually for each participant. Randomization will be performed using computer-generated random sequences (randomizer.org), with predefined randomization sets created prior to study initiation.

Each position will be maintained for approximately 5 minutes. In each position, end-expiratory lung impedance difference (ΔEELI) will be measured using the upright sitting position as the reference. The total duration of the study protocol is expected to be approximately 30 minutes per participant. The study will be completed once all measurements have been obtained in all positions.

ELIGIBILITY:
Inclusion Criteria:

-BMI between 18-25 kg/m² or 30-40 kg/m²

Exclusion Criteria:

* Individuals with a body mass index (BMI) between 25 and 30 kg/m²,
* Pregnancy
* Respiratory tract infection within the previous two weeks
* Anatomical abnormalities of the chest wall that may interfere with Electrical Impedance Tomography (EIT) measurements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy non-obese and obese volunteers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
MI | Periprocedural
  Match Index (MI, 0-100%): quantifying the spatial overlap of ventilation and perfusion distributions. MI values will be taken from the device's Match View. Change in Match Index (MI) between obese and non-obese participants across positions will be compared.

SECONDARY OUTCOMES:
VV % | Periprocedural
  Percentage of ventral ventilation across body positions.
DV % | Periprocedural
  Percentage of dorsal ventilation across body positions.
VP % | Periprocedural
  Percentage of ventral perfusion across body positions.
DP % | Periprocedural
  Percentage of dorsal perfusion across body positions.
DI % | Periprocedural
  Dead space index (DI), proportion (in %) of lung units (pixels or ROIs) that are ventilated but not perfused across body positions
SI % | Periprocedural
  Shunt index (SI), proportion (in %) of lung units (pixels or ROIs) that are perfused but not ventilated across body positions
GI | Periprocedural
  Global Inhomogeneity Index (0-100) quantifies how evenly ventilation is distributed across the lung regions. Higher values indicate more heterogeneous ventilation distribution across the lung cross-section.
CoV | Periprocedural
  Center of ventilation (CoV) describes the center of mass of the ventilation distribution along the ventrodorsal axis (0-100, from ventral to dorsal). CoV <40% means more ventral ventilation while >50-55% means more dorsal ventilation.
ΔEELI | Periprocedural
  ΔEELI represents the change in end-expiratory lung impedance measured by EIT between each body position and the upright sitting reference position, reflecting relative changes in end-expiratory lung volume associated with positioning.
Heart rate | Periprocedural
  Heart rate per minute measured by pulse oximetry
Oxygen saturation | Periprocedural
  Oxygen saturation measured by pulse oximetry

CONTACTS AND LOCATIONS:
Overall Officials: Evren Şentürk, MD, Study Director — Koç University School of Medicine
Locations (1):
- Koç University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data collected for the study, including de-identified individual participant data will be made available to other within 6 months after the publication of this trial, as will additional related documents (study protocol, statistical analysis plan and informed consent form), for academic purposes (e.g , meta-analyses) upon request to the corresponding author, and with a signed data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after the publication
Access Criteria: Academic purposes

REFERENCES:
- [Background] De Jong A, Wrigge H, Hedenstierna G, Gattinoni L, Chiumello D, Frat JP, Ball L, Schetz M, Pickkers P, Jaber S. How to ventilate obese patients in the ICU. Intensive Care Med. 2020 Dec;46(12):2423-2435. doi: 10.1007/s00134-020-06286-x. Epub 2020 Oct 23. PMID 33095284